CLINICAL TRIAL: NCT05082792
Title: The Role of Doppler Ultrasound in Assessment of Local Factors Affecting Maturation of Arteriovenous Fistula in Hemodialysis Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Areej Mahmoud Ibrahim, Resident doctor at diagnostic and interventional radiology department Sohag University Hospitals, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-21-10-21
Record Dates: First submitted 2021-10-15; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Doppler Ultrasound in Arteriovenous Fistula Preoperative Evaluation and Post-operative Periodic Monitoring
Keywords: hemodialysis in CKD. AVF. CDUS
MeSH Terms: interventions — Ultrasonography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- doppler US for native AVF in upper limb (Other): creation of native arteriovenous fistula in upper limb in chronic kidney disease patients on hemodialysis
  Interventions: Diagnostic Test: doppler ultrasound

INTERVENTIONS:
Diagnostic Test: doppler ultrasound — Doppler ultrasound evaluation of AVF:
  * pre-operative evaluation: venous system (patency of central veins and deep venous system, patency of superficial veins, the latter diameter, depth form skin surface, distance from nearby artery, any sizable adjacent tributaries), and arterial system including morphological evaluation (course, diameter, wall alterations, any stenoocclusive disorders) and functional evaluation (flow volume and ability to dilate)
  * post-operative evaluation: anastomotic site (type of anastomosis, patency, diameter, PSV and any other morphologic alterations), inflow afferent artery (diameter, PSV and flow volume), outflow efferent vein (patency, diameter, color flow, spectral waveform)
  * the first post-operative sonographic evaluation will be done after removal of stiches from the wound and periodic monitoring every one week up until completion of 6 weeks

SUMMARY:
the long term survival of the chronic kidney disease (CKD) patients depends on the adequacy of dialysis via good vascular access. the arteriovenous fistula (AVF) is the preferred vascular access for hemodialysis. pre-operative evaluation and periodic monitoring of the AVF after creation with well-defined applied criteria by color doppler ultrasound (CDUS) will help to reduce rate of access failure and achieve better cumulative patency rate of fistulas.

DETAILED DESCRIPTION:
In recent years, the improvement in the diagnosis and treatment of chronic kidney disease (CKD) has led to increase the number of patients who need hemodialysis, adequacy of which depends upon the appropriately placed vascular access. Although the arteriovenous fistula (AVF) is the preferred vascular access for hemodialysis, there is still a high rate of failure to mature in clinical practice. To increase the use of AVFs, especially in the co-morbid patients, a thorough pre-operative evaluation and periodic monitoring after AVF creation by color doppler ultrasound (CDUS) allows placement of AVF in higher proportion of patients, and early detection of access dysfunction with subsequent intervention that reduce the rate of access failure.

Doppler ultrasound is the main imaging modality for assessment of dialysis access circuits as its gives information on the morphological criteria and evaluates the inflow and outflow flows. CDUS is non-invasive modality, of low cost, not using ionizing radiation or iodinated contrast media.

ELIGIBILITY:
Inclusion Criteria:

CKD and ESRD patients on hemodialysis, in whom native arteriovenous fistula operation is needed

* both sexes are included.
* age group from 15-80years
* upper limb arteriovenous fistula only.
* native arteriovenous fistula.
* surgically succeeded AVF

Exclusion Criteria:

we will exclude:

* patients refused to be in the research.
* Patients with AVF not in the upper limbs.
* Patient of age less than 15years and above 80years.
* patients with synthetic grafts.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
maturation of AVF | 6 months
  maturation is considered successful if the fistula patent has a diameter >6mm, located <6mm maximum depth from skin surface, with PSV 400cm/s, flow volume 600ml/min, within 6 weeks post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

REFERENCES:
- [Background] 1. Malekmakan L, Haghpanah S, Pakfetrat M et al (2009) Causes of chronic renal failure among Iranian hemodialysis patients. Saudi J Kidney Dis Transpl. 20(3):501-504 2. Shaheen AMFA, Al-Khader A (2005) Epidemiology and causes of end stage renal disease (ESRD). Saudi J Kidney Dis Transplant. 16(3):277-281 3. Malovrh M (2005) Native arteriovenous fistula: preoperative evaluation. Am J Kidney Dis. 39:1218-1225 4. Yerdel MA, Kesenci M, Yazicioglu KM et al (1997) Effect of hemodynamic variables on surgically created arteriovenous fistula flow. Nephrol Dial Transplant. 12(8):1684-1688 5. Wilmink T, Hollingworth L, Powers S et al (2016) Natural history of common autologous arteriovenous fistulae: consequences for planning of dialysis access. Eur J Vasc Endovasc Surg. 51:134-140 6. Lee T (2013) Novel paradigms for dialysis vascular access: downstream vascular biology-is there a final common pathway? Clin J Am Soc Nephrol. 8:2194-2201